CLINICAL TRIAL: NCT02470559
Title: Treatment of High Risk or Recurrent Ovarian Cancer With Anti-CD3 x Anti-HER2 Bispecific Antibody Armed Activated T Cells (BATs), Low Dose IL-2, and GM-CSF (Phase I).
Brief Title: Activated T-cell Therapy, Low-Dose Aldesleukin, and Sargramostim in Treating Patients With Ovarian, Fallopian Tube, or Primary Peritoneal Cancer That is Stage III-IV, Refractory, or Recurrent
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study did not accrue any participants, the PI has left the institution.
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Lawrence Lum, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-129; NCI-2015-00180 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-129 (Other: Barbara Ann Karmanos Cancer Institute); P30CA022453 (NIH)
Record Dates: First submitted 2015-06-10; First posted 2015-06-12 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Malignant Ovarian Clear Cell Tumor; Malignant Ovarian Serous Tumor; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma; Stage IIIA Fallopian Tube Cancer; Stage IIIA Ovarian Cancer; Stage IIIA Primary Peritoneal Cancer; Stage IIIB Fallopian Tube Cancer; Stage IIIB Ovarian Cancer; Stage IIIB Primary Peritoneal Cancer; Stage IIIC Fallopian Tube Cancer; Stage IIIC Ovarian Cancer; Stage IIIC Primary Peritoneal Cancer; Stage IV Fallopian Tube Cancer; Stage IV Ovarian Cancer; Stage IV Primary Peritoneal Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — aldesleukin; sargramostim; Colony-Stimulating Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (aldesleukin, sargramostim, HER2Bi-aACT) (Experimental): Patients receive HER2Bi-aATC IV over 5-15 minutes and IP within 3-4 days of IV dose weekly for 4 weeks. Patients also receive low-dose aldesleukin SC daily and sargramostim SC twice weekly beginning 3 days before the first HER2Bi-aATC infusions infusion and ending 7 days after the last HER2Bi-aATC infusion. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Aldesleukin; Biological: HER2Bi-Armed Activated T Cells; Other: Laboratory Biomarker Analysis; Biological: Sargramostim

INTERVENTIONS:
Biological: Aldesleukin — Given SC
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; Recombinant Human Interleukin-2
Biological: HER2Bi-Armed Activated T Cells — Given IV and IP
  Other Names: Anti-CD3 x Anti-Her2/neu Bispecific Antibody-Armed Activated T Cells; HER2Bi-Armed ATCs
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Sargramostim — Given SC
  Other Names: 23-L-Leucinecolony-Stimulating Factor 2; DRG-0012; Leukine; Prokine; rhu GM-CFS; Sagramostim; Sargramostatin

SUMMARY:
This phase I trial studies the side effects and best dose of activated T-cell therapy when given together with low-dose aldesleukin and sargramostim in treating patients with ovarian, fallopian tube, or primary peritoneal cancer that is stage III-IV, has not responded to previous treatment, or has come back. Activated T cells that have been coated with bi-specific antibodies, such as anti-cluster of differentiation (CD)3 and anti-human epidermal growth factor receptor 2 (HER2), may stimulate the immune system in different ways and stop tumor cells from growing. Aldesleukin may stimulate white blood cells to kill tumor cells. Colony-stimulating factors, such as sargramostim, may increase the production of blood cells. Giving activated T-cell therapy with low-dose aldesleukin and sargramostim may be a better treatment for ovarian, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Perform a phase I clinical trial consisting of dose-escalation/de-escalation of intraperitoneal (IP) infusions of anti-CD3 x anti-HER2/neu (HER2Bi) armed anti-CD3 activated T cells (aATC) in women with high risk or recurrent ovarian cancer to determine the maximum tolerated dose (MTD) for IP injections in combination with a fixed intravenous (IV) dose of 10 x 10^9 (± 20%) aATC once a week.

II. To clearly define the toxicity profile of IP and IV HER2Bi aATC at the MTD or technically feasible dose in patients with ovarian cancer.

SECONDARY OBJECTIVES:

I. Evaluate clinical responses, time to progression, and overall survival. II. Evaluate phenotype, cytokine profiles and interferon (IFN)-gamma enzyme-linked immunosorbent spots (ELISPOTS), cytotoxicity and antibodies directed at laboratory ovarian cancer cell lines.

III. Monitor cancer antigen (CA)125 or tumor markers, and antibody responses to mouse proteins (human anti-mouse antibodies [HAMA]).

IV. The migration of armed ATC out of the peritoneal and serum cytokine levels induced by IP or IV armed ATC infusion will be assessed by studying the appearance of armed ATC at various time points (0, 4, 8, 12, 24, 48, 72, and 96 hours after IP infusion) in the blood after IP infusions by performing flow cytometry to detect anti-CD3 (OKT3) x anti-Her2 (Herceptin®) bi-specific antibody (BiAb) on the surface of aATC.

OUTLINE: This is a dose-escalation study of IP infused HER2Bi-armed activated T cells.

Patients receive HER2Bi-aATC IV over 5-15 minutes and IP within 3-4 days of IV dose weekly for 4 weeks. Patients also receive low-dose aldesleukin subcutaneously (SC) daily and sargramostim SC twice weekly beginning 3 days before the first HER2Bi-aATC infusions infusion and ending 7 days after the last HER2Bi-aATC infusion. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 1 and 3 months, and then every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented, epithelial ovarian, fallopian tube, or primary peritoneal, high grade serous or clear cell carcinoma are eligible; all patients must have a confirmed pathology; stage 3 and 4 initial disease with response to primary surgery and neo/adjuvant chemotherapy, platinum refractory disease, and patients with recurrent disease are candidates
* Patients meeting the above pathologic criteria will be eligible for therapy irrespective of their HER2/neu over expression status; immunohistochemical staining will be not be required for protocol entry but fluorescence in situ hybridization (FISH) and immunohistochemistry (IHC) studies for HER2/neu are preferred
* Chemotherapy: no limit to prior therapies; however, patients with multiple chemotherapy regimens will be screened for lymphocyte proliferation at investigator's discretion
* Herceptin: women who have been previously treated with Herceptin or other monoclonal antibody therapies are eligible for the trial
* Radiation therapy: patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis are excluded; prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients may have no evidence of measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria or have measurable disease; CA-125 and other available markers will be obtained
* Karnofsky performance score of >= 70 is required or Eastern Cooperative Oncology Group (ECOG) score, performance status (PS) = 0-2
* The patient must have a life expectancy of 3 months or more based on the judgment of the investigators; women who have rapidly progressive symptomatic disease affecting major organ systems such as the liver and lungs will be excluded
* Negative serum test for pregnancy in premenopausal women
* No previous or concurrent malignancy, other than curatively treated in situ squamous cell carcinoma of the cervix or basal cell carcinoma of the skin or non-active breast cancer
* Each patient must be aware of the nature of her disease process and must willingly consent to treatment after being informed of alternatives, potential benefits, side effects, and risks; eligibility testing that is considered standard of care may be done prior to informed consent but no immunotherapy related procedures or testing may occur without informed consent
* No serious medical or psychiatric illness which prevents informed consent or intensive treatment
* Patients will be ineligible for treatment on this protocol if:

  * There is a history of a recent myocardial infarction (within one year)
  * There is a history of a past myocardial infarction (more than one year ago) along with current coronary symptoms requiring medications and/or evidence of depressed left ventricular function (left ventricular ejection fraction [LVEF] < 45% by echocardiogram [ECHO])
  * There is a current history of angina/coronary symptoms requiring medications and/or evidence of depressed left ventricular function (LVEF < 45% by ECHO)
  * There is clinical evidence of congestive heart failure requiring medical management (irrespective of ECHO results)
* Patients who have persistently elevated systolic blood pressures (BPs) >= 145 or diastolic BPs >= 90 need to have their systolic or diastolic BP controlled with anti-hypertensive agents for at least 3 days prior to the initiation of cell therapy; patients already on anti-hypertensive agents will have their medicine adjusted based on the clinical judgment of the patient care team
* Patients with treated brain metastases (received definitive radiation and/or underwent surgical resection) are eligible for therapy on this protocol; patients with clinical evidence of active brain metastases are ineligible for therapy on this protocol
* Granulocytes >= 1,000/mm^3
* Platelet count >= 50,000/ul
* Hemoglobin >= 8 gm/dl
* Blood urea nitrogen (BUN) =< 1.5 times normal
* Serum creatinine =< 1.8 mg/dl
* Creatinine clearance >= 60 ml/mm
* Bilirubin =< 2.0 times normal
* Serum glutamic oxaloacetic transaminase (SGOT) =< 2.0 times normal
* Human immunodeficiency virus (HIV) = negative
* LVEF >= 45% at rest (by ECHO)
* Pulmonary function tests (PFT)-forced expiratory volume in one second (FEV1), diffusing capacity of the lung for carbon monoxide (DLCO2), and forced vital capacity (FVC) >= 60% predicted value if clinically indicated
* Minor changes from the required initial laboratory data guidelines will be allowed at the discretion of the attending team under special circumstances; the reasons for exceptions must be documented prior to enrollment
* Appropriate slides of the primary lesion will be available for future review; if available, HER2/neu positivity will be recorded
* Peritoneal dialysis catheter implantation is identical to that from the Gynecologic Oncology Group (GOG) 252 Protocol and revised from the GOG Surgical Procedures Manual

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
MTD of IP injections in combination with the IV fixed dose of aATC determined by the incidence of dose-limiting toxicity (DLT) defined using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0 | Up to 4 weeks
Toxicity profile of IP and IV HER2Bi-aATC at the MTD or technically feasible dose graded using NCI CTCAE version 4.0 | Up to 2 years
  Patients who received any armed ATC but not evaluable for DLT will be analyzed separately for the toxicity profile. The toxicity will be summarized with point and exact confidence intervals.

SECONDARY OUTCOMES:
Changes in cytokine profiles | Baseline to up to 12 months
  Increases or decreases in the amount of cytokine produced from the pre immunotherapy baseline at any time point after immunotherapy will be considered as continuous outcomes. Paired t-test or Wilcoxon signed rank test will be used to compare the difference between baseline and after any time point of aATC treatment in proliferation, ELISPOTS, and the amount of cytokine produced. The data collected at all study time points after immunotherapy will be analyzed using mixed-effect model for longitudinal data adjusted for baseline measures.
Changes in HAMA levels in serum samples | Baseline to up to 12 months
  Sera from patients will be obtained before and after immunotherapy at the designated time points to determine if there is development of HAMA responses directed at OKT3 (mouse IgG2a antibody). Paired t-test or Wilcoxon signed rank test will be used to compare the difference between baseline and after any time point of aATC treatment in proliferation, ELISPOTS, and the amount of cytokine produced. The data collected at all study time points after immunotherapy will be analyzed using mixed-effect model for longitudinal data adjusted for baseline measures.
Changes in phenotyping induced by immunotherapy in peripheral blood mononuclear cells (PBMC) | Baseline to up to 12 months
  PBMC from the patients will be obtained before and after immunotherapy to determine if there changes induced by immunotherapy. Paired t-test or Wilcoxon signed rank test will be used to compare the difference between baseline and after any time point of aATC treatment in proliferation, ELISPOTS, and the amount of cytokine produced. The data collected at all study time points after immunotherapy will be analyzed using mixed-effect model for longitudinal data adjusted for baseline measures.
Clinical response rate (including complete response, partial response, progressive disease, and stable disease) measured on the basis of CA-125 or RECIST-defined tumor measurements | Up to 12 months
  Point and exact confidence interval estimates will be calculated for response rate.
Increases in IFN-gamma ELISPOTS | Baseline to up to 12 months
  Paired t-test or Wilcoxon signed rank test will be used to compare the difference between baseline and after any time point of aATC treatment in proliferation, ELISPOTS, and the amount of cytokine produced. The data collected at all study time points after immunotherapy will be analyzed using mixed-effect model for longitudinal data adjusted for baseline measures.
Increases in the immunoglobulin G titer against selected ovarian cancer cell lines in serum samples | Baseline to 4 weeks
  Sera from patients will be obtained before and after immunotherapy to determine if there are changes induced by immunotherapy. Paired t-test or Wilcoxon signed rank test will be used to compare the difference between baseline and after any time point of aATC treatment in proliferation, ELISPOTS, and the amount of cytokine produced. The data collected at all study time points after immunotherapy will be analyzed using mixed-effect model for longitudinal data adjusted for baseline measures.
Overall survival | From the beginning of immunotherapy to the time of death, assessed up to 12 months
  Will be estimated with the standard Kaplan-Meier method, from which summary statistics of interest (median, 6 month, 1-year rate, etc.) will be derived. Both point and 95% confidence interval estimates will be calculated.
Progression free survival | From the beginning of immunotherapy to progression or death, assessed up to 12 months
  Will be estimated with the standard Kaplan-Meier method, from which summary statistics of interest (median, 6 month, 1-year rate, etc.) will be derived. Both point and 95% confidence interval estimates will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Lum, Principal Investigator — Barbara Ann Karmanos Cancer Institute